CLINICAL TRIAL: NCT01011946
Title: Staging of Axillary Lymph Nodes Using the PEM Flex Solo II Pet Scanner in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 16893A
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Positron Emission Mammography (Experimental)
  Interventions: Device: Positron Emission Mammography

INTERVENTIONS:
Device: Positron Emission Mammography — Patients will receive bilateral (both sides) breast and axillary PEM scans, bilateral mammography, DCE-MRI, US of the breast and axilla (the side of the affected breast), and ultrasound guided biopsy of axillary lymph node if suspicious. Various PEM views will be performed on both your breast and axilla (underarm).

SUMMARY:
The purpose of this study is to determine if PEM scan can improve axillary lymph node staging by assessing if they are involved by cancer. Your doctor may refer you for a PEM scan, PEM stands for positron emission mammography, a relatively new and advanced application of positron emission tomography or PET scanning. For decades, PET has helped doctors diagnose and treat disease.

DETAILED DESCRIPTION:
Subjects will receive bilateral (both sides) breast and axillary PEM scans. All recruited subjects chosen for the study will have biopsy proven breast cancer and are eligible for chemotherapy. They will undergo bilateral breast MRI for staging which is considered standard of care. Breast MRI and PEM scans will be performed at at baseline (phase 0 or pre-operative phase), 2nd MRI and PEM after 1 to 2 weeks of NAC (phase 1) and 3rd MRI and PEM after 1 to 2 weeks of phase 1 (phase 2). DCE-MRI and PEM will be performed not more than 14 days apart within each phase. Cranio-Caudal (CC) and Medial Lateral Oblique (MLO) PEM views will be performed of both the ipsilateral and contralateral breast and axillae by a Mammography Technologist trained in mammographic positioning.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-75 years old with newly diagnosed breast cancer who are considered candidates for breast conserving surgery (i.e. lumpectomy).

Exclusion Criteria:

* Children (<18 years old)
* Pregnant or Lactating women
* Diabetic patients (Type I or II)
* Patients who are scheduled for a sentinel node procedure using radioactive Tc-99m within 24 hours of PEM
* Patients who have NOT undergone a standard of care bilateral breast MRI at UC.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Appelbaum, M.D., Principal Investigator — The University of Chicago Medical Center
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positron Emission Mammography
Started | 36
Completed | 33
Not Completed | 3
Not completed — Transferred to another hospital | 2
Not completed — No pathological lab value | 1

BASELINE CHARACTERISTICS:
Arm/Group | Positron Emission Mammography
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of FDG Positron Emission Mammography (PEM) in Identifying Axillary Lymph Node (ALN) Metastases From Breast Cancer
Description: Based on FDG Positron Emission Mammography (PEM) image, a breast region was classified as "normal" or "abnormal". Lymph Node (LN) sampling and histopathology determined true positives and true negatives.
Time Frame: PEM was performed prior to surgery and LN sampling immediately following surgery
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Positron Emission Mammography
Number analyzed (Participants) | 33
percentage of subjects
  Sensitivity | 83.3 [51.6 to 97.9]
  Specificity | 52.0 [31.3 to 72.2]

ADVERSE EVENTS:
Arm/Group | Positron Emission Mammography
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes